CLINICAL TRIAL: NCT06541080
Title: Collection of Liquid Biopsy Samples of Patients With Neuroendocrine Neoplasms - CollectNET 2.0, a Study by the BE-FORCE Consortium
Brief Title: Collection of Liquid Biopsy Samples of Neuroendocrine Neoplasms (NEN) Patients - Collection of NET (CollectNET) 2.0, a Study by the BE-FORCE Consortium
Acronym: BE-FORCE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Universiteit Antwerpen (Other); KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: B3002021000275
Record Dates: First submitted 2024-07-11; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-12

CONDITIONS: Neuroendocrine Neoplasms
Keywords: liquid biopsy; circulating cell-free DNA; methylation-based biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regular Sampling Group (RSG): This group consists of all NEN patients who have measurable tumor burden on imaging (and who do not fulfill the criteria for the Intensive Sampling Group) and are willing to participate in the study.
  Interventions: Diagnostic Test: Shallow Whole Genome Sequencing (sWGS)-GIPXplore; Diagnostic Test: methylation-sensitive restriction enzymes (MSRE)-Single-molecule molecular inversion probes (smMIP)-seq assay
- Intensive Sampling Group (ISG): This group consists of patients who at baseline or during the course of the study patients in this group (i) have a histologically confirmed NEN of WHO 2019 grade 1-3 NET or NEC from pancreatic, colorectal, or small intestinal origin and (ii) are starting any kind of 1st line systemic treatment (e.g. somatostatin analogues, targeted therapy, chemotherapy, etc.).
  Interventions: Diagnostic Test: Shallow Whole Genome Sequencing (sWGS)-GIPXplore; Diagnostic Test: methylation-sensitive restriction enzymes (MSRE)-Single-molecule molecular inversion probes (smMIP)-seq assay

INTERVENTIONS:
Diagnostic Test: Shallow Whole Genome Sequencing (sWGS)-GIPXplore — GIPXplore will be used to mine shallow whole genome sequencing cell free DNA data for identification of signatures.
Diagnostic Test: methylation-sensitive restriction enzymes (MSRE)-Single-molecule molecular inversion probes (smMIP)-seq assay — Aberrant methylation in ccfDNA will be analyzed using the novel, highly sensitive MSRE-smMIP-seq technology.

SUMMARY:
The CollectNET 2.0 by BE-FORCE is a prospective, multicentric, interventional study in which liquid biopsies will be collected from neuroendocrine neoplasms (NEN) patients to create an extensive biobank that will be used for current and future circulating cell-free DNA (ccfDNA) analyses. Two sampling groups will be created: the "Regular Sampling Group" and the "Intensive Sampling Group". Upon participation, up to four additional blood tubes (max. total of 32.5mL) will be collected at each timepoint as specified below. These include 3 Streck Cell-Free DNA tubes (10 mL each) which will be used for the extraction of ccfDNA and 1 PreAnalytiX (PAXgene)® Blood RNA tube (2.5 mL). All NEN patients in one of the participating hospitals who have measurable tumor burden on imaging will be asked to participate in our study and will be included in the "Regular Sampling Group". If additionally, the patient is (i) diagnosed with a histologically confirmed NEN of World Health Organisation (WHO) 2019 grade 1-3 neuroendocrine tumor (NET) or neuroendocrine carcinoma (NEC) from pancreatic, colorectal or small intestinal origin and (ii) is starting any kind of 1st line systemic treatment (e.g. somatostatin analogues, targeted therapy, chemotherapy, etc.), they will be followed up more intensively as per the "Intensive Sampling Group". If during follow-up in this "Intensive Sampling Group" patients have disease progression or have completed follow-up for 3 years in this group, their follow-up will switch back to the "Regular Sampling Group" for the remainder of the study. Ultimately, the samples collected in the "Intensive Sampling Group" will be used to achieve the second and third objective of our current project. These are to validate novel ccfDNA analyzing techniques (IMPRESS and GIPXplore) for assessment of the presence and quantification of circular tumor DNA (ctDNA) in liquid biopsies, and to monitor tumor fraction (i.e., ctDNA quantities) over time in sequential plasma samples from NEN patients using ccfDNA assays and correlating this with time to progression (according to RECIST 1.1 criteria) to explore the predictive efficacy of ccfDNA analysis and thereby evaluate its biomarker potential for patient follow-up. While samples from the "Regular Sampling Group" and the PAXgene tubes will be biobanked for future projects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age on the day of signing informed consent.
* Written informed consent must be obtained from the patient or patient's legal representative.
* Patient is willing and able (in the investigator's opinion) to comply with all trial requirements.
* For inclusion in the Regular Sampling Group: patients must have (had) a histologically confirmed NEN diagnosis, patients must have measurable tumor burden on imaging, patients must be in follow-up in one of the participating hospitals and patients who have progressed or completed follow-up for 3y in the Intensive Sampling Group.
* For inclusion in the Intensive Sampling Group: patients who are included in the Regular Sampling Group and where either a baseline sample (RSG-B) or a recent RSG follow-up sample (RSG-V…) has been collected before the start of 1st systemic treatment (as defined below), patients must be diagnosed with a histologically confirmed NEN diagnosis of a WHO 2019 grade 1-3 NET or NEC of pancreatic, colorectal, or small intestinal origin and patients must start any kind of 1st line systemic treatment (e.g. somatostatin analogues, targeted therapy, chemotherapy, etc.).

Exclusion Criteria:

* Patients who are unable to give informed consent.
* Patients for which blood sampling would compromise their overall health.
* Patients pregnant at time of study entry or are willing to become pregnant during the study.
* Patients with a history or current evidence of any condition or abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NEN patients
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2028-12-04 (Estimated); Study Completion 2030-12-04 (Estimated)

PRIMARY OUTCOMES:
Validating novel ccfDNA analyzing techniques for assessment of the presence and quantification of ctDNA in liquid biopsies derived from NEN patients | 5 years after informed consent form (ICF) signature
  ctDNA fraction
Monitoring tumor fraction over time in sequential plasma samples from NEN patients using ccfDNA assays | 5 years after ICF signature
  ctDNA quantities
Correlate tumor fraction with time to progression (according to RECIST 1.1 criteria) | 5 years after ICF signature
  tumor fraction

CONTACTS AND LOCATIONS:
Overall Officials: Timon Vandamme, Principal Investigator — University Hospital, Antwerp
Locations (8):
- Belgium (8):
  - AZ Rivierenland, Rumst, Antwerp
  - VITAZ, Sint-Niklaas, East-Flanders
  - University Hospital Leuven, Leuven, Flemish Brabant
  - Ziekenhuis Netwerk Antwerpen (ZNA), Antwerp
  - Gasthuiszusters Ziekenhuizen (GZA), Antwerp
  - AZ Monica, Antwerp
  - AZ Klina, Brasschaat
  - Antwerp University Hospital (UZA), Edegem

IPD SHARING:
Plan to Share IPD: No